CLINICAL TRIAL: NCT04502017
Title: Efficacy of Different Anti-Thrombotic Strategies on Device-Related Thrombosis Prevention After Percutaneous Left Atrial Appendage Occlusion
Acronym: FADE-DRT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Texas Cardiac Arrhythmia Research Foundation (Other)
Responsible Party: Principal Investigator, Andrea Natale, Executive Medical Director, Texas Cardiac Arrhythmia Research Foundation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TCAI_LAAO
Record Dates: First submitted 2020-08-04; First posted 2020-08-06 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Device-Related Thrombosis; Atrial Fibrillation; Left Atrial Appendage Occlusion
Keywords: left atrial appendage; Watchman; antithrombotic therapy; device-related thrombosis
MeSH Terms: conditions — Atrial Fibrillation | interventions — Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Antithrombotic Therapy (Active Comparator): OAC for 6 weeks followed by DAPT until 6 month-follow-up, then aspirin alone
  Interventions: Drug: ASA plus Clopidogrel
- Genetic-Tailored AntiThrombotic Strategy (Active Comparator): OAC for 6 weeks followed by DAPT (clopidogrel responders) or aspirin plus half-dose OAC (clopidogrel non-responders) until 6 month-follow-up, then aspirin alone
  Interventions: Drug: Genetic-Tailored AntiThrombotic Strategy
- Half-Dose NOAC (Active Comparator): Half Dose of Novel OAC
  Interventions: Drug: Half-Dose of novel OAC

INTERVENTIONS:
Drug: ASA plus Clopidogrel — OAC (6 weeks) + DAPT (until 6 months) + ASA
  Arms: Standard Antithrombotic Therapy
Drug: Genetic-Tailored AntiThrombotic Strategy — Half-Dose OAC or Clopidogrel in combination with ASA on the basis of CYP2C19 Genotype
  Arms: Genetic-Tailored AntiThrombotic Strategy
Drug: Half-Dose of novel OAC — Half Dose of novel OAC post-device Implantation
  Arms: Half-Dose NOAC

SUMMARY:
Comparison among three different antithrombotic strategies after percutaneous LAA occlusion with a Watchman FLX LAAC device.

DETAILED DESCRIPTION:
Data on the optimal antithrombotic therapy (AT) after percutaneous left atrial appendage (LAA) occlusion are still scarce. The classical AT strategy after LAA occlusion includes 6-weeks of warfarin + aspirin followed by dual anti platelet therapy with clopidogrel (75 mg) and aspirin (81-325 mg) until 6 months of follow-up, then aspirin alone is continued indefinitely. Nonetheless, a significant number of patients continues to suffer from device-related thrombosis which carries a high risk of thromboembolic events. Other AT strategies have been tested in order to reduce the risk of thrombus-formation on device. Among them, replacement of clopidogrel with half-dose oral anticoagulation (OAC) in patients with genetic resistance to this drug has been recently reported to reduce the incidence of DRT. Additionally, reduced dose of novel OAC was demonstrated to lead to lower thrombin generation compared to DAPT.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥18 years of age
* Successful LAAC procedure (device implanted without procedural or bleeding complication).
* Patients contraindicated or unsuitable for long-term OAC.
* History of AF (permanent or persistent or paroxysmal).
* Written informed consent by the patient or designee if the patient is unable to consent

Exclusion Criteria:

* Life expectancy < 2 years.
* Pregnant, breastfeeding, or unwilling to practice birth control during participation in the study.
* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2020-08-05 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Composite of Stroke, Systemic Embolism, and Device-related Thrombosis | 1 year
Incidence of Major Bleeding Events | 1 year

SECONDARY OUTCOMES:
Incidence of Minor Bleeding Events | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- St. David's Medical Center, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No